CLINICAL TRIAL: NCT05647915
Title: Assess the Effects of Berberine in Reducing Abdominal Visceral Adipose Tissue Among Individuals with Obesity and Non-alcoholic Fatty Liver Disease
Brief Title: Effects of Berberine in Reducing Abdominal Visceral Adipose Tissue Among Individuals with Obesity and NAFLD
Acronym: BRAVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-CXGC04-2
Record Dates: First submitted 2022-11-16; First posted 2022-12-13 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Obesity, Abdominal; NAFLD
Keywords: berberine hydrochloride
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Non-alcoholic Fatty Liver Disease | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data manager and statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- berberine group (Experimental): Berberine hydrochloride plus lifestyle intervention
  Interventions: Drug: Berberine plus lifestyle intervention
- placebo group (Placebo Comparator): Placebo plus lifestyle intervention
  Interventions: Behavioral: Placebo plus lifestyle intervention

INTERVENTIONS:
Drug: Berberine plus lifestyle intervention — berberine hydrochloride 500mg twice a day for 6 months plus lifestyle intervention.
  Lifestyle intervention is based on "Guidelines of prevention and treatment for non-alcoholic fatty liver disease (2018 update)" and "China Blue Paper on Obesity Prevention and Control", including health education on diet, physical activity and weight loss, etc.
  Arms: berberine group
Behavioral: Placebo plus lifestyle intervention — Placebo with identical shape, colour, odour and taste twice a day plus lifestyle intervention.
  Lifestyle intervention is based on "Guidelines of prevention and treatment for non-alcoholic fatty liver disease (2018 update)" and "China Blue Paper on Obesity Prevention and Control", including health education on diet, physical activity and weight loss, etc.
  Arms: placebo group

SUMMARY:
This multicenter, double-blinded, randomized controlled trial aims to evaluate the effect of berberine in reducing visceral and liver adipose tissue among individuals with obesity and non-alcoholic fatty liver disease (NAFLD) in China.

DETAILED DESCRIPTION:
The trial aims to evaluate the efficacy and safety of berberine treatment for obesity and NAFLD. Potential eligible patients will be recruited from 10-20 medical centers in China. After a 4-week run-in period with berberine, all the eligible participants will be randomized (1:1) to berberine 1.0 g per day plus lifestyle intervention (Arm A) or placebo plus lifestyle intervention (Arm B). The participants will be asked to attend the visit at least once every 2 months, and be followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 years
* Participants with obesity (i.e., BMI ≥ 28 kg/m2) and abdominal obesity (i.e., waist circumference ≥85 cm in female or waist circumference ≥90 cm in male)
* Participants with NAFLD diagnosed by ultrasound, computed tomography or magnetic resonance imaging

Exclusion Criteria:

* Patients with established coronary heart disease, stroke, or peripheral arterial disease
* Patients diagnosed with diabetes or taking oral glucose-lowering drugs
* Patients with severely uncontrolled hypertension (i.e., SBP≥180mmHg and/or DBP ≥110mmHg)
* Excess alcohol consumption (i.e., alcohol ≥ 20 g/day in female or alcohol ≥ 30 g/day in male)
* Other causes of fatty liver disease, including alcohol or drug abuse, hepatitis B or C, autoimmune, hepatolenticular degeneration, total parenteral nutrition, inflammatory bowel disease, celiac disease, hypothyroidism, Cushing syndrome, β -lipoprotein deficiency, lipid atrophy diabetes, Mauriac syndrome, etc.
* Patients with thyroid disease, including hyperthyroidism or hypothyroidism
* Patients with cardiac insufficiency
* ALT or AST ≥ 3 times upper limit of normal, liver cirrhosis or hepatic insufficiency
* Patients with renal insufficiency: estimated glomerular filtration rate (eGFR) < 60 ml/(min×1.73m2)
* Patients who had weight loss surgery, or are currently taking drugs for weight loss, or plan to have weight loss surgery or drugs in the following 6 months
* Patients diagnosed with glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Taking berberine or drug containing berberine in the past 1 month
* Any adverse reaction to berberine
* Severe constipation, diarrhea, and/or severe chronic intestinal diseases (e.g., ulcerative colitis, Crohn's disease, irritable bowel syndrome, etc.)
* Patients who had to use long-term or intermittent corticosteroids, immunosuppressants, antibiotics, or other drugs that affect inflammatory biomarkers
* Women who are pregnant or breastfeeding, or those who plan to be pregnant during the trial
* Patients with malignant tumors
* Patients with mental disorders, cognitive disorders, and/or other serious diseases
* Those who participated or have been participating other trials during the last 3 months
* Any other conditions that may hinder the compliance to the study intervention or follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Change of visceral fat content | 6 months
  Measurement of visceral fat by computed tomography
Change of liver fat content | 6 months
  Measurement of liver fat content by computed tomography

SECONDARY OUTCOMES:
Change of fasting plasma glucose | 6 months
  Measurement of fasting plasma glucose (FPG)
Change of HbA1c | 6 months
  Measurement of HbA1c
Change of 2-hour postprandial blood glucose | 6 months
  Measurement of 2-hour postprandial blood glucose (2hPG)
Change of homeostatic model assessment-insulin resistance | 6 months
  Homeostatic model assessment-insulin resistance (HOMA-IR)= (fasting insulin (mIU/L) * FPG (mmol/L)) / 22.5
Change of homeostasis model assessment-β cell | 6 months
  Homeostatic model assessment (HOMA-β) = (20 x fasting insulin (mIU/L)) / (FPG (mmol/L) - 3.5)
Change of homeostasis model assessment-insulin sensitivity | 6 months
  Homeostatic model assessment-insulin sensitivity (HOMA-IS)= 1/ HOMA-IR
Change of serum triglyceride | 6 months
  Measurement of serum triglyceride (TG)
Change of high-density lipoprotein cholesterol | 6 months
  Measurement of high-density lipoprotein cholesterol
Change of low-density lipoprotein cholesterol | 6 months
  Measurement of low-density lipoprotein cholesterol
Change of total cholesterol | 6 months
  Measurement of total cholesterol
Change of lipoprotein (a) | 6 months
  Measurement of lipoprotein (a)
Change of apolipoprotein | 6 months
  Measurement of apolipoprotein
Normalization of glucose parameters among participants with prediabetes | 6 months
  Meeting all three criteria: 1) FPG<6.1 mmol/L; 2) 2hPG<7.8 mmol/L; 3) HbA1c<5.7%
Change of metabolic syndrome z-score | 6 months
  Metabolic syndrome z-score calculated by the five components, including waist circumference, HDL-C, blood pressure, TG and FPG. Higher score indicates greater severity of metabolic syndrome
Change of visceral fat index | 6 months
  Visceral fat index calculated by waist circumference, body mass index, TG, HDL-C. Higher index indicates higher content of visceral fat
Change of fat liver index | 6 months
  Fat liver index (FLI) calculated by TG, body mass index, gamma-glutamyltransferase (γ-GGT), waist circumference. Higher index indicates higher content of liver fat
Change of triglyceride glucose index | 6 months
  Triglyceride glucose index (TyG) calculated by TG and FPG. Higher index indicates higher insulin resistance
Change of serum urine acid | 6 months
  Measurement of serum urine acid
Change of serum homocysteine | 6 months
  Measurement of serum homocysteine
Change of body weight | 6 months
  Measurement of body weight in kg
Change of body mass index | 6 months
  Weight and height will be combined to report BMI in kg/m^2
Change of waist circumference | 6 months
  Measurement of waist circumference in cm
Change of waist-hip ratio | 6 months
  Waist circumference and hip circumference will be combined to report waist-hip ratio.
Change of waist-height ratio | 6 months
  Waist circumference and height will be combined to report waist-height ratio.
Change of systolic blood pressure | 6 months
  Measurement of systolic blood pressure (SBP)
Change of diastolic blood pressure | 6 months
  Measurement of diastolic blood pressure (DBP)

OTHER OUTCOMES:
Change of alanine aminotransferase | 6 months
  Measurement of alanine aminotransferase (ALT)
Change of aspartate aminotransferase | 6 months
  Measurement of aspartate aminotransferase (AST)
Change of γ-GGT | 6 months
  Measurement of γ-GGT
Change of fibrosis-4 score | 6 months
  Fibrosis-4 score (FIB-4) calculated by age, ALT, AST, platelet count. Higher score indicates higher extent of liver fibrosis.
Change of NAFLD fibrosis score | 6 months
  NAFLD fibrosis score (NFS) calculated by age, BMI, status of dysglycemia, ALT, AST, platelet count, serum albumin concentration. Higher score indicates higher extent of liver fibrosis.
Change of hypersensitive C-reactive protein | 6 months
  Measurement of hypersensitive C-reactive protein
Change of interleukin-6 | 6 months
  Measurement of interleukin-6 (IL-6)
Change of tumor necrosis factor-α | 6 months
  Measurement of tumor necrosis factor-α (TNF-α)
Change of transforming growth factor-β | 6 months
  Measurement of transforming growth factor-β (TGF-β)
Change of leptin | 6 months
  Measurement of leptin
Change of adiponectin | 6 months
  Measurement of adiponectin
Change of short chain fatty acids | 6 months
  Measurement of short chain fatty acids
Change of trimethylamine | 6 months
  Measurement of trimethylamine (TMA)
Change of trimethylamine oxide | 6 months
  Measurement of trimethylamine oxide (TMAO)
Improvement of left ventricular diastolic function (LVDF) among participants with abnormal LVDF at baseline | 6 months
  Measurement of LVDF by echocardiogram
Change of pericardial fat among participants with abnormal LVDF | 6 months
  Measurement of pericardial fat by computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, PhD, Principal Investigator — National Center for Cardiovascular Diseases; Haibo Zhang, MD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, National Center for Cardiovascular Diseases, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan HM, Xia MF, Wang Y, Chang XX, Yao XZ, Rao SX, Zeng MS, Tu YF, Feng R, Jia WP, Liu J, Deng W, Jiang JD, Gao X. Efficacy of Berberine in Patients with Non-Alcoholic Fatty Liver Disease. PLoS One. 2015 Aug 7;10(8):e0134172. doi: 10.1371/journal.pone.0134172. eCollection 2015. PMID 26252777
- [Background] Harrison SA, Gunn N, Neff GW, Kohli A, Liu L, Flyer A, Goldkind L, Di Bisceglie AM. A phase 2, proof of concept, randomised controlled trial of berberine ursodeoxycholate in patients with presumed non-alcoholic steatohepatitis and type 2 diabetes. Nat Commun. 2021 Sep 17;12(1):5503. doi: 10.1038/s41467-021-25701-5. PMID 34535644
- [Derived] Lei L, Wang B, Zhao L, Li J, Yan X, Jiang J, Wang L, Ren G, Li Y, Cheng X, Yan X, Zhu Y, Guo Y, Zhong H, Zhang H, Li J; BRAVO Collaborative Group. Berberine and Adiposity in Diabetes-Free Individuals With Obesity and MASLD: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2554152. doi: 10.1001/jamanetworkopen.2025.54152. PMID 41543854